CLINICAL TRIAL: NCT01016028
Title: Chemotherapy-Induced Peripheral Neuropathy: Feasibility and Validity of New Symptom Measurement Tools in Patients on Treatment With Platinum Agents, Taxanes and Bortezomib
Brief Title: Chemotherapy-Induced Peripheral Neuropathy Survey
Status: Withdrawn | Type: Observational
Why Stopped: Study assessment tool development delayed.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0439
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer; Colorectal Cancer; Myeloma; Chemotherapy-induced Peripheral Neuropathy
Keywords: Cancer; Colorectum Cancer; Colorectal disease; neuropathic symptom tool; chemotherapy-induced peripheral neuropathy; CIPN; Pain; Quantitative Sensory Testing; QST; symptom measurement tools; platinum agents; cisplatin; oxaliplatin; taxanes; bortezomib
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Neoplasms, Plasma Cell; Neoplasms; Pain | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire + Sensory Tests + Interview
  Interventions: Behavioral: Questionnaire; Behavioral: Sensory Tests; Behavioral: Interview

INTERVENTIONS:
Behavioral: Questionnaire — 3 questionnaires to collect information about any pain and/or symptoms experienced, general well-being, and personal information such as age and marital status. One (1) will be a symptom assessment questionnaire where asked to rate symptoms on a scale of 0-10.
  Other Names: Survey
Behavioral: Sensory Tests — Test of sensitivity to things such as cold and touch, involve feeling cold objects, feeling bumps on a rectangular board, and putting pegs into holes on a board; and marking on computerized drawings areas experience pain, numbness, and/or cold sensitivity.
Behavioral: Interview — First 5 patients receiving platinum agents, taxanes, and bortezomib (15 patients total) will be asked to describe their symptoms in an open-ended, semi-structured 20-30 minute interview.

SUMMARY:
The goal of this research study is to learn more about pain and other symptoms that patients may experience while receiving chemotherapy treatment with platinum agents, taxanes, and/or bortezomib.

DETAILED DESCRIPTION:
If patient agrees to take part in this study, they will be asked to complete 3 questionnaires, 3 sensory tests, and may be asked to take part in a one-on-one symptom interview.

Symptom Interview:

Depending on when patient is enrolled in this study, they may take part in a one-on-one interview with a study staff member. A total of 15 participants will take part in this interview (5 taking platinum agents, 5 taking taxanes, & 5 taking bortezomib). During the interview, patient will be asked to describe their symptoms. The interview should take about 20-30 minutes to complete.

The interviews will be digitally recorded, transcribed (typed), and used by researchers to identify symptoms related to receiving this type of chemotherapy. Researchers will use this information to design a study questionnaire that focuses on chemotherapy symptoms in the hands and feet. The digital recordings and typed copies of the interview will be destroyed after researchers have analyzed the interview data and the study is complete.

Questionnaires & Sensory Tests:

All study participants will complete 3 questionnaires that are designed to collect information about any pain and/or symptoms patient may have experienced, their general well-being, and personal information such as age and marital status. One (1) of them is called a symptom assessment questionnaire and patient be will asked to rate their symptoms on a scale of 0-10.

All study participants will also complete 3 tests, called sensory tests, that are designed to help researchers learn how sensitive patient is to things such as cold and touch. These tests involve feeling cold objects, feeling bumps on a rectangular board, and putting pegs into holes on a board. Patient will also be asked to mark on computerized drawings the areas where they experience any pain, numbness, and/or cold sensitivity. A study staff member will explain how to take the tests and use the computerized drawings in more detail at the time these tests are performed.

It should take about 20-30 minutes to complete all of the questionnaires and tests.

Additional Sensory Testing:

Out of the 200 participants on this study, 40 participants will be asked to return to the clinic for additional sensory testing to help researchers learn if the tools used for this study are working as expected.

This additional testing is designed to help researchers learn how sensitive patient is to things such as touch, cold, warmth, and a pinprick to the finger, hand, or arm. Patient will be asked to describe how well they can feel each test, and how much pain they may or may not feel. This additional testing should take about 60 minutes to complete.

Length of Study:

After patient has completed the interview (if they are asked), 3 questionnaires, and 3 sensory tests their participation on this study will be over. If patient is selected to take part in the additional sensory testing, their participation on this study will be over after those tests are complete.

This is an investigational study.

Up to 200 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >= 18 years old.
2. Patients must be fluent with the English language.
3. Patients must be on chemotherapy regimes with any of the study drugs: cisplatin, oxaliplatin, taxanes and/or bortezomib.

Exclusion Criteria:

1. Significant cognitive impairment as determined by the trained research staff
2. Chronic alcoholism or substance abuse
3. Diagnosis of severe depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, age 18 years or older, receiving chemotherapy with cisplatin or oxaliplatin (platinum agents), taxanes, and/or bortezomib at UT MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Assessment of Patient's Symptoms (Questionnaire) | Each patient administered questionnaire at single point in time.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cleeland, PHD,BA, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org